CLINICAL TRIAL: NCT06849661
Title: Do Preoperative Bilirubin Levels Affect Recovery and Hospital Stay After Sedation Anesthesia?
Status: Enrolling by invitation | Type: Observational
Sponsor: Naime Yalçın (Other)
Responsible Party: Sponsor-Investigator, Naime Yalçın, Specialist Anesthesiology and Reanimation, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: KAEK/2025.01.4
Record Dates: First submitted 2025-02-15; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Preoperative Biliary Drainage; Recovery Period, Anesthesia; Hospital Length of Stay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Bilirubines (Total,direct,indirect), Amylase, AST, ALT, ALP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arm Low Bilirubine Levels
- Arm High Bilirubine Levels

SUMMARY:
There are still complexities regarding the effects of anesthetic drugs on bilirubin metabolism. The aim of the study was to investigate whether preoperative serum bilirubin levels are associated with the length of hospital stay after ERCP performed under sedation anesthesia in the presence of propofol. Unstable hemodynamics, increased propofol sensitivity, and prolonged recovery time to anesthetics are common features encountered in patients with hyperbilirubinemia. Therefore, close monitoring of cardiovascular functions in these patients and awareness of the possible need for a reduction in the dose of anesthetic used are the expected benefits of the study.

DETAILED DESCRIPTION:
Bilirubin is a lipid-soluble substance produced as the end product of heme metabolism in mammals. It easily crosses cell membranes, including the blood-brain barrier (BBB), and has been reported to have both neuroprotective and neurotoxic effects. Most bilirubin binds to albumin, but unbound bilirubin crosses the BBB, binds to nerve cells, and exhibits cytotoxic effects. Neurological symptoms resulting from hyperbilirubinemia are common in neonates, but decrease after BBB maturation. However, patients may be susceptible/vulnerable to neurological complications as a result of liver cirrhosis, decreased albumin production, or drug-induced displacement of bilirubin from albumin binding sites. It can also cause a blood-brain barrier dysfunction in situations such as anesthesia/surgery. In addition to playing a protective role, bilirubin also plays a role in the progression of neurological dysfunction in many pathological conditions. Many of these conditions elevate bilirubin concentrations above physiological levels, where the toxic effects of bilirubin begin to outweigh its protective antioxidant benefits and damage the nervous system. Bilirubin becomes neurotoxic when it reaches micromolar concentrations, the same level at which it aggregates and adheres to cell membranes, disrupting normal cell function. High bilirubin levels, or hyperbilirubinemia, are classically defined as bilirubin levels greater than 3 mg/dL and should typically be considered a sign of an underlying disease state. Jaundice is often a symptom of underlying liver and biliary tract disease. Hyperbilirubinemia most often refers to liver/biliary tract disease, but it can be the result of a variety of hereditary causes or can also be caused by hematologic disorders. Endoscopic retrograde cholangiopancreatography (ERCP) was initially developed in 1968 as an important diagnostic tool for biliary and pancreatic diseases. Patients were injected with a dye and referred to an interventional radiologist or a surgeon for further treatment if necessary. Dr. William S. McCune performed the first successful ERCP using a fiber duodenoscope. In 1972, Dr. Peter Cotton described cannulation in 60 patients. The following year, Dr. Meinhard Classen in Germany and Dr. Keiichi Kawai in Japan simultaneously performed the first biliary sphincterotomy. ERCP has moved from being a diagnostic tool to a therapeutic tool. The complication and mortality rates associated with ERCP have been reported as 5% to 10% and 0.1% to 1%, respectively. It is a complex and time-consuming procedure that can be performed with deep sedation or general anesthesia. There is no consensus on the best anesthetic application between deep sedation and general anesthesia. While benzodiazepines and opioids have traditionally been used for sedation, propofol has recently become popular worldwide. Propofol has a rapid onset and end of action, and its hypnotic properties provide patient comfort and amnesia. This ultimately leads to faster recovery and increased ERCP success and satisfaction. Complications such as respiratory depression and hypoxemia are observed in association with sedation, with a frequency ranging from 2% to 26%. The incidence is directly proportional to the duration of the procedure, and the odds ratio increases from 1.8 in procedures lasting less than 10 minutes to 7.9 in procedures lasting more than 1 hour. The ability of drugs used in anesthesia to remove bilirubin from albumin has not been studied adequately. There is no specific data on the protein binding of propofol, but it is known that propofol removes bilirubin induced by fatty acid components from albumin, causing an increase in free bilirubin. However, one study indicated that the concentration of unconjugated bilirubin is generally relatively small and that the effect of propofol on albumin binding is insignificant. It was stated that the main issue to be considered is the possible effects of this large number of conjugated bilirubins on propofol binding. It was stated that conjugated bilirubin is water soluble and the two propofol regions in human serum albumin are hydrophobic; therefore, it is unlikely that conjugated bilirubin will compete with propofol at these sites. Another study has suggested that although bilirubin levels do not change the free concentration of propofol, the free concentration of propofol may increase significantly if the human serum albumin concentration in these patients with impaired liver function falls significantly.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* ASA I-IV status
* Both genders
* To be operated under sedation anesthesia for ERCP procedure

Exclusion Criteria:

* age <18
* pregnancy
* lack of informed consent (such as patients with mental retardation or
* language problems)
* history of allergy to any agent used during sedation
* baseline O2 saturation <90%
* baseline systolic blood pressure <90 mmHg
* procedure performed under general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on patients who applied to the anesthesia polyclinic of SBU University Kanuni Sultan Süleyman E.A.H. and were scheduled to undergo ERCP under sedation. A total of 360 patients over the age of 18, ASA I-IV status, of both genders, who will undergo an ERCP procedure under sedation anesthesia will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative bilirubin levels and length of hospital stay | from the beginning of the enrollment until 1 month after sedation anesthesia recovery
  Patients' age, gender, weight in kilograms, height in centimeter, weight and height will be combined to report BMI in kg/m^2, chronic disease history, medication history, smoking, alcohol, ASA status, being an inpatient or outpatient, Hb (hemoglobin), platelets, Na (sodium), K (potassium), INR (international normalized ratio), total bilirubin, direct bilirubin, indirect bilirubin, ALP (Alkaline phosphatase), ALT (Alanine aminotransferase), AST (aspartate aminotransferase), and hospital stay will be recorded by reviewing the case follow-up forms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)